CLINICAL TRIAL: NCT06656156
Title: Effects of Proprioceptive Neuromuscular Facilitation of Iliopsoas and Hamstring on Patients With Chronic Low Back Pain
Brief Title: PNF Technique on Iliopsoas and Hamstring Muscle on Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01944 Aisha
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain
Keywords: Low back pain; Proprioceptive neuromuscular facilitation (PNF); Mechanical; Chronic pain; Iliopsoas and hamstring
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive neuromuscular facilitation technique (Experimental): Proprioceptive neuromuscular facilitation technique along with conventional treatment
  Interventions: Other: Proprioceptive neuromuscular facilitation technique
- Conventional treatment (Active Comparator): Tens and hotpack
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation technique — Experimental group was given proprioceptive neuromuscular facilitation technique (PNF) along with conventional treatment.
  PNF will be applied on iliopsoas and hamstring muscles, 3 repetitions/session with a break of 2 minutes/repetition (10 second isometric Contraction then 10 second stretch)
  Treatment contains total 12 sessions (3 times/week for 4 consecutive weeks)
  Arms: Proprioceptive neuromuscular facilitation technique
Other: Conventional treatment — Conventional treatment contains tens and hotpack.
  Tens Will be applied for 20 minutes and hotpack for 10 minutes
  Total 12 sessions (3 times/week for 4 consecutive weeks)
  Arms: Conventional treatment

SUMMARY:
The aim of the study to evaluate the effects of PNF in terms of decreasing low back pain, increasing range of motion and improving flexibility of the hamstrings and iliopsoas. Their association in LBP can be found through studies and my study based on this point will show whether targeting these two muscles would have any effect on lumbar back pain.

DETAILED DESCRIPTION:
One of the most prevalent, significant, and leading causes of disability in industries is chronic low back pain (CLBP) which also leads to poor quality of life. 50.4% of patients with low back pain reported a history of prolonged unsupported sitting. A study which evaluates muscle tightness in women desk job workers shows 89.83% have Hamstring tightness, whereas 35.59% have Iliopsoas tightness. In today's world majority of jobs require long hours sitting or standing with limited body movements like those involving computers and visual displays, bankers, teachers, industrial workers, architects, and so forth. This sedentary lifestyle has a negative effect on muscles, leads to the shortening which was one of the main contributors to the development of LBP. The iliopsoas, along with other back muscles, is said to play an essential role in stabilizing the pelvis. the shortening of the iliopsoas muscle produced inappropriate loading on the lumbar spine, mostly resulting in greater lumbar lordosis and anterior pelvic tilting thereby acting as a risk factor for low back pain. Patients with LBP also reported shorting of hamstring muscles due to Long-duration sitting.

When treating low back pain, physiotherapy is just as helpful as medication. For acute, chronic, or subacute low back pain, take into consideration the addition of non-pharmacological therapy that has been shown to be beneficial. PNF technique is one of the specific advanced physical exercises.

Joint movement limitation, traction, stretching, and resisted movement are all part of proprioceptive neuromuscular facilitation (PNF). It is effective for restoring ROM, strength, and flexibility to injured or stiff muscles. The PNF Method depends on movement patterns that enhance sensory-motor function. It has been proposed that PNF corrects the distorted impulses generated from muscle proprioceptive receptors. As a result, it lessens discomfort and aims to increase muscle strength.

Proprioceptive neuromuscular facilitation (PNF) is a form of flexibility exercises used to resolve muscle shortening and straining. Studies show that PNF stretching can help individuals with chronic back pain by improving hip range of motion, functional impairment, and pain management. According to a literature review published from 1970 to February 2020, PNF was more effective in helping people suffering with chronic low back pain to relieve their pain and enhance their waist function. A study of India, in 2015 concluded that PNF (modified hold relax) was more effective than ART at increasing hamstring flexibility and reducing pain and impairment. A study conducted in 2017 shows, PNF(CRAC) stretching technique on iliopsoas combined with hamstring stretching is effective to reduce back pain. In just one session, the PNF group had experienced significantly more benefits than the MET group in terms of pain relief, lumbar lordosis reduction, and loosening of the tight iliopsoas. A thesis comparing between PNF exercise and McKenzie method, in which PNF exercise shows better improvement in the low back pain than McKenzie method. another study supports the literature that when treating patients with chronic low back pain, the rhythmic stabilization training technique of proprioceptive neuromuscular facilitation combined with a series of isotonic exercises proved to be beneficial than either technique used alone. Researchers also observed that application of PNF stretching significantly reduces low back pain and dysfunction in patients with chronic low back pain.

In a study they have analyzed the relationship between the iliopsoas and hamstring tightness on LBP. The most powerful and deep hip flexor is the iliopsoas muscle, which is not normally stretched during daily activities. People whose occupations require them to sit for extended periods of time may notice a shortening of these muscles due to adaptation changes. Tightness in that area causes anterior pelvic tilting and hyper-lordosis of the spine, which strain the back muscles and eventually results in low back pain. Muscle flexibility increases and the pelvis retrovert and neutralize when we stretch the iliopsoas. A study found an association between passive hip extension and prolonged sitting/physical inactivity. Results showed there was 6.1° more passive hip extension in the high activity & minimal sitting group when compared to the low activity & prolonged sitting group. muscle imbalances due to muscle tension and weakness affects neutral lumbopelvic alignment, among them hamstring extensibility is considered the most important. The tightness in the hamstring causes the adaptive shortening of the muscles leading to posterior pelvic tilt along with the flattening of the lumbar spine which causes pain in the low back. A study concluded that Participants with low back pain had significantly shorter hamstring muscle length than participants without low back pain. Moreover, the hamstring is one of the stabilizers of the pelvic motion in the sagittal plane by controlling the anterior pelvic tilt.

When iliopsoas muscle shortens, the hip joint's biomechanics get disrupted to cause anterior pelvic tilting, according to literature in order to compensate iliopsoas tightness, hamstring contracts to hold the pelvis in its position, which can lead to its tightness because of constant remaining in contracted phase and vice versa. this pathophysiology affects the lumber spine's curvature and causes low back discomfort and exaggeration of subjective symptoms. PNF stretching improves mobility and helps in the healing of injuries by using reflexes to produce deeper stretches that loosen up tight muscles.

The aim of the study to evaluate the effects of PNF in terms of decreasing low back pain, increasing range of motion and improving flexibility of the hamstrings and iliopsoas. Their association in LBP can be found through studies and my study based on this point will show whether targeting these two muscles would have any effect on lumbar back pain. And as there is no published literature available in national evidence on the effects of the PNF technique on either hamstring or iliopsoas tightness, my study bridges the gap and will be a beneficial addition to the literature and also will recommend a cost-effective, easy and harmless treatment that can be implemented as an effective treatment for low-back pain patients.

ELIGIBILITY:
Inclusion Criteria:

* chronic NSLBP of more than 3 months (NPRS 3-7)
* positive modified Thomas test (Posterior thigh does not touch table, knee flex >80)
* positive modified SLR (unable to extend knee), SLR (pain >70 degrees)

Exclusion Criteria:

* History of abdominal, back, and hip surgery
* Spine and hip fracture
* menstruation at the time of testing.
* Pain and severe joint stiffness of hip and knee
* problems of cardiovascular and respiratory systems
* Physiological problems that cause referred pain at the low back (UTI, kidney problem, tumor, pancreatitis)
* Pregnancy

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale( NPRS) | 4th week
  Changes from baseline Numeric pain rating scale starting from 0 to 10 (0-3 categories as mild, 4-6 as moderate and 7-10 as severe) used to assess pain of lumber spine

SECONDARY OUTCOMES:
ROM lumber spine flexion | 4th week
  Changes from baseline ROM (range of motion) of lumber spine flexion will be taken with the help of Goniometer
ROM lumber spine extension | 4th week
  Changes from baseline ROM (range of motion) of lumber spine extension will be taken with the help of Goniometer
ROM lumber spine side bend | 4th week
  Changes from baseline ROM (range of motion) of lumber spine side bend will be taken with the help of Goniometer
ROM lumber spine rotation | 4th week
  Changes from baseline ROM (range of motion) of lumber spine rotation will be taken with the help of Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: shamaila yaqub, Ms-ompt, Principal Investigator — Riphah International University
Locations (1):
- Jinnah postgraduate Medical centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lakkadsha TM, Qureshi MI, Kovela RK, Saifee SS, Lalwani SS. Efficacy of Single Stretching Session of Iliopsoas Using Proprioceptive Neuromuscular Facilitation Versus Muscle Energy Technique on Low Back Pain in Patients With Lumbar Hyper-Lordosis. Cureus. 2022 Aug 12;14(8):e27916. doi: 10.7759/cureus.27916. eCollection 2022 Aug. PMID 36110466
- [Background] Gao P, Tang F, Liu W, Mo Y. The effects of proprioceptive neuromuscular facilitation in treating chronic low back pain: A systematic review and meta-analysis. J Back Musculoskelet Rehabil. 2022;35(1):21-33. doi: 10.3233/BMR-200306. PMID 34250930
- [Background] Cejudo A, Centenera-Centenera JM, Santonja-Medina F. The Potential Role of Hamstring Extensibility on Sagittal Pelvic Tilt, Sagittal Spinal Curves and Recurrent Low Back Pain in Team Sports Players: A Gender Perspective Analysis. Int J Environ Res Public Health. 2021 Aug 16;18(16):8654. doi: 10.3390/ijerph18168654. PMID 34444402